CLINICAL TRIAL: NCT05459675
Title: Effects of Very Low-calorie Diet Versus Bariatric Surgery on Body Composition and Gut Microbiota Pattern in Obese Patients
Brief Title: Effects of Very Low-calorie Diet Versus Bariatric Surgery on Body Composition and Gut Microbiota Pattern
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chanawit Saiyalam, Faculty of Medicine Ramathibodi Hospital Mahidol University, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MURA2016/647
Record Dates: First submitted 2022-06-02; First posted 2022-07-15 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: Very low-calorie diet; Bariatric surgery; Body composition; Gut microbiota pattern
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Three groups of patients will be recruited at obesity clinic, Ramathibodi Hospital Mahidol University, Bangkok, Thailand. One group will take part in the very low-calorie diet (VLCD). One group will be undergone bariatric surgery (LRYGB or LSG)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very low-calorie diet (Experimental): Patients in the very low-calorie diet group will be prescribed a very low-calorie diet (meal replacement) for 12 weeks, then the patients will be monitored up to 1 year
  Interventions: Other: Very low-calorie diet
- Bariatric surgery (Experimental): Patients in the bariatric surgery group will be undergone bariatric surgery LRYGB and will be follow-up according the current guideline
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Other: Very low-calorie diet — Meal replacement (800 kcal/day, protein 90 g/day)
  Arms: Very low-calorie diet
Procedure: Bariatric surgery — Bariatric surgery will be performed by single surgeon at Ramathibodi Hospital Mahidol University, Thailand. Postoperative diet progression according to the current guideline will be prescribed from early post-op period to 1 year after surgery
  Arms: Bariatric surgery

SUMMARY:
Obesity is a chronic disease characterized by the excessive accumulation of fat in body and it continues to be a major public health problem worldwide. Treatment options for obesity include lifestyle modification, pharmacotherapy and bariatric surgery. Bariatric surgery is a highly effective treatment for obesity and results in rapid and sustained weight loss. Also, it significantly alters gut microbiota composition and function. A very low-calorie diet (VLCD) is a rapid weight loss program which calorie intake is severely restricted (< 800 kcal/day). It has been shown to be very effective to induce rapid weight loss and result in comorbidities resolution similar to bariatric surgery. Therefore, this study was aimed to study the effects of 12-week VLCD compare to bariatric surgery (Laparoscopic Roux-en-Y gastric bypass (LRYGB) or Laparoscopic Sleeve Gastrectomy (LSG)) on weight loss, body composition, gut microbiota pattern and other metabolic parameters.

DETAILED DESCRIPTION:
The study will include obese patients (body mass index; BMI ≥ 37.5 kg/m2 or BMI ≥ 32.5 kg/m2 with comorbidities), aged 15-65 years at Ramathibodi Hospital, Thailand. The VLCD group will received total diet replacement for 12 weeks and the bariatric surgery group will undergo LRYGB or LSG. Study participants in both groups will be matched according to their age, sex, body mass index (BMI) and diabetic status. Body weight reduction and body composition, gut microbiota pattern, liver stiffness and steatosis, glycemic and other metabolic parameters (glucose, insulin, c-peptide, lipid profile, liver function test, kidney function test, complete blood count, electrolyte blood test, thyroid function tests, serum ketone and adiponectin), health-related quality of life, depression score and twenty-four-hour diet recall and physical activity will be assessed at baseline and at month 1, 3, 6, 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-65 years
* Male or female
* Body mass index ≥ 32.5 kg/m2 with obesity related co-morbidity
* Body mass index ≥ 37.5 kg/m2 with or without an obesity related co-morbidity

Exclusion Criteria:

* End stage disease such as cancer, cirrhosis Child-Pugh C, critical/acute illness
* Type 1 diabetes mellitus
* Recent eGFR < 30 ml/min/1.73 m2
* Weight loss ≥ 5% in the previous 3 months
* Use of antibiotics in the previous 1 month
* Use of probiotic or prebiotic supplement in form of tablet or sachet in the previous 14 days
* Current treatment with anti-obesity drugs
* Pregnancy or breast feeding
* Substance abuse
* Uncontrolled psychiatric disorder and eating order
* History of allergy to any components in meal replacement product or whey protein product
* Unable to give informed consent

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | From baseline to 12 weeks
  Weight in kg

SECONDARY OUTCOMES:
Body Composition | From baseline to 12 weeks
  The percentage of body fat and skeleton muscle mass
Gut microbiota pattern | From baseline to 12 weeks
  Measured by 16S ribosomal RNA (rRNA) gene sequencing on the fecal samples
Liver stiffness | From baseline to 12 weeks
  Measured by FibroScan® instrument
Liver steatosis | From baseline to 12 weeks
  Measured by FibroScan® instrument
Blood pressure | From baseline to 12 weeks
  Systolic and diastolic blood pressure
Fasting plasma glucose | From baseline to 12 weeks
  Measured in mg/dl
Hemoglobin A1c | From baseline to 12 weeks
  Measured in %
Fasting insulin | From baseline to 12 weeks
  Measured in μIU/l
Insulin resistance | From baseline to 12 weeks
  Measured by the homeostatic model of insulin resistance (HOMA-IR)
Triglyceride | From baseline to 12 weeks
  Measured in mg/dl
Total cholesterol | From baseline to 12 weeks
  Measured in mg/dl
LDL-cholesterol | From baseline to 12 weeks
  Measured in mg/dl
HDL-cholesterol | From baseline to 12 weeks
  Measured in mg/dl
Health-related quality of life | From baseline to 12 weeks
  Measured by the EQ-5D-5L questionnaire
Depression | From baseline to 12 weeks
  Measured by the PHQ-9 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wharton S, Lau DCW, Vallis M, Sharma AM, Biertho L, Campbell-Scherer D, Adamo K, Alberga A, Bell R, Boule N, Boyling E, Brown J, Calam B, Clarke C, Crowshoe L, Divalentino D, Forhan M, Freedhoff Y, Gagner M, Glazer S, Grand C, Green M, Hahn M, Hawa R, Henderson R, Hong D, Hung P, Janssen I, Jacklin K, Johnson-Stoklossa C, Kemp A, Kirk S, Kuk J, Langlois MF, Lear S, McInnes A, Macklin D, Naji L, Manjoo P, Morin MP, Nerenberg K, Patton I, Pedersen S, Pereira L, Piccinini-Vallis H, Poddar M, Poirier P, Prud'homme D, Salas XR, Rueda-Clausen C, Russell-Mayhew S, Shiau J, Sherifali D, Sievenpiper J, Sockalingam S, Taylor V, Toth E, Twells L, Tytus R, Walji S, Walker L, Wicklum S. Obesity in adults: a clinical practice guideline. CMAJ. 2020 Aug 4;192(31):E875-E891. doi: 10.1503/cmaj.191707. No abstract available. PMID 32753461
- [Background] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Background] Scheithauer TPM, Rampanelli E, Nieuwdorp M, Vallance BA, Verchere CB, van Raalte DH, Herrema H. Gut Microbiota as a Trigger for Metabolic Inflammation in Obesity and Type 2 Diabetes. Front Immunol. 2020 Oct 16;11:571731. doi: 10.3389/fimmu.2020.571731. eCollection 2020. PMID 33178196
- [Background] Shao Y, Ding R, Xu B, Hua R, Shen Q, He K, Yao Q. Alterations of Gut Microbiota After Roux-en-Y Gastric Bypass and Sleeve Gastrectomy in Sprague-Dawley Rats. Obes Surg. 2017 Feb;27(2):295-302. doi: 10.1007/s11695-016-2297-7. PMID 27440168
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Umphonsathien M, Prutanopajai P, Aiam-O-Ran J, Thararoop T, Karin A, Kanjanapha C, Jiamjarasrangsi W, Khovidhunkit W. Immediate and long-term effects of a very-low-calorie diet on diabetes remission and glycemic control in obese Thai patients with type 2 diabetes mellitus. Food Sci Nutr. 2019 Feb 11;7(3):1113-1122. doi: 10.1002/fsn3.956. eCollection 2019 Mar. PMID 30918654
- [Background] Lane M, Howland G, West M, Hockey M, Marx W, Loughman A, O'Hely M, Jacka F, Rocks T. The effect of ultra-processed very low-energy diets on gut microbiota and metabolic outcomes in individuals with obesity: A systematic literature review. Obes Res Clin Pract. 2020 May-Jun;14(3):197-204. doi: 10.1016/j.orcp.2020.04.006. Epub 2020 Jun 13. PMID 32546361
- [Background] Guo Y, Huang ZP, Liu CQ, Qi L, Sheng Y, Zou DJ. Modulation of the gut microbiome: a systematic review of the effect of bariatric surgery. Eur J Endocrinol. 2018 Jan;178(1):43-56. doi: 10.1530/EJE-17-0403. Epub 2017 Sep 15. PMID 28916564
- [Background] Damms-Machado A, Mitra S, Schollenberger AE, Kramer KM, Meile T, Konigsrainer A, Huson DH, Bischoff SC. Effects of surgical and dietary weight loss therapy for obesity on gut microbiota composition and nutrient absorption. Biomed Res Int. 2015;2015:806248. doi: 10.1155/2015/806248. Epub 2015 Feb 1. PMID 25710027
- [Background] Castaner O, Goday A, Park YM, Lee SH, Magkos F, Shiow STE, Schroder H. The Gut Microbiome Profile in Obesity: A Systematic Review. Int J Endocrinol. 2018 Mar 22;2018:4095789. doi: 10.1155/2018/4095789. eCollection 2018. PMID 29849617